CLINICAL TRIAL: NCT06782984
Title: Patient-derived Organoids As Predictive Models for Drug Response Testing and Repurporsing in Glioblastoma Therapy
Brief Title: Drug Response Testing and Repurposing Using Glioblastoma Organoid
Status: Recruiting | Type: Observational
Sponsor: Chungnam National University Hospital (Other)
Collaborators: Korea Advanced Institute of Science and Technology (Other); Keimyung University Dongsan Medical Center (Other); Soonchunhyang University Hospital (Other); Dong-A University Hospital (Other); Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Kyung Hwan Kim, Assistant Professor, Chungnam National University Hospital
Other Study IDs: CNUH 2021-08-020-012
Record Dates: First submitted 2025-01-06; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma; Organoid
Keywords: organoid; glioblastoma; GBO; drug-screening
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — tumor tissues and organoids
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- glioblastoma: prospectively enrolled
  Interventions: Other: Organoid-based drug sensitivity test

INTERVENTIONS:
Other: Organoid-based drug sensitivity test — The intervention in this study involves utilizing glioblastoma organoids (GBOs) to perform an organoid-based drug sensitivity test (DST) and retrospectively comparing the results with clinical outcomes. Notably, no interventions will be applied to participants based on GBO-DST results; the study is limited to retrospective analysis.
  The GBO-DST is conducted by performing a drug response assay with temozolomide to determine the half-maximal inhibitory concentration (IC50), which serves to classify GBOs as TMZ-sensitive or TMZ-resistant. This classification is further validated through GBO cell survival analysis.

SUMMARY:
The aim of this observational study, based on a prospectively collected cohort, is to evaluate the prognostic value of patient-derived organoids in predicting responses to conventional and repurposing drugs, including temozolomide, in patients with primary or recurrent glioblastoma. The primary question is whether the patient's response to temozolomide is recapitulated in their corresponding patient-derived glioblastoma organoid (GBO). Patient drug responses are evaluated using survival data, while GBO drug responses are assessed through a drug-response testing platform utilizing cell viability assays. Additionally, this platform is used to explore the potential application of various chemotherapeutic agents.

DETAILED DESCRIPTION:
Glioblastoma multiforme (GBM) remains a highly aggressive brain tumor with limited treatment options and a poor prognosis. Temozolomide (TMZ) is the only approved first-line therapy, but frequent resistance limits its efficacy, highlighting the urgent need for alternative treatments. Patient-derived glioblastoma organoids (GBOs) offer a promising preclinical model for personalized drug testing and therapy development.

In our previous study, we established 20 GBO lines using a serum-free protocol, preserving the histopathological and genomic features of the parental tumors. Additionally, GBO Drug Sensitivity Testing (GBO-DST) was developed to evaluate TMZ responsiveness and to screen several FDA-approved drugs, including Lazertinib and Regorafenib. The GBO-DST was successfully validated by correlating IC50 values with progression-free survival, GBO size measurement after treatment, and histopathological evaluation.

The goal of this study is to investigate whether a preclinical model using GBOs can eventually replace clinical trials. Therefore, it is necessary to collect diverse genetic information from patients in a multicenter setting, along with corresponding GBOs that recapitulate the patient tumors. Using GBO-DST, external cohort validation will be performed. Concurrently, the study aims to predict the potency of multi-kinase inhibitors or EGFR-TKIs, which are expected to show efficacy based on prior research, and compare these predictions against clinical outcomes.

This study aims to establish 100 GBO lines, targeting the enrollment of 150 patients, considering a previous success rate of 66.7% for GBO establishment. Since the study requires tumor tissue and genetic information from patients, IRB approvals from multiple institutions have been secured (including five tertiary hospitals in South Korea: Chungnam National University Hospital, Soonchunhyang University Hospital, Keimyung University Hospital, Yeungnam University Hospital, and Dong-A University Hospital). However, as this study retrospectively correlates patient clinical outcomes with GBO-DST results, it does not involve direct interventions with patients. Specifically, GBO-DST results for multiple candidate drugs will not be used to alter patients' treatment regimens.

The study collects clinical information and genetic data from patients, with clinical outcomes defined as progression-free survival and overall survival. Radiologic data will be prospectively collected to achieve these objectives.

Through this study, we aim to validate the findings of previous research by confirming that GBO-DST accurately recapitulates patients' drug responses. Furthermore, we seek to establish GBO-DST as a preclinical trial platform capable of replacing traditional clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* primary or recurrent glioblastoma
* patients treated with standard treatment including surgery and temozolomide based chemoradiation therapy
* sufficient tumor sample is available for organoid culture

Exclusion Criteria:

* patients who are not underwent concurrent chemoradiation therapy (CCRT) following surgery
* failed to obtain MRI scan after CCRT
* patients refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with primary or recurrent glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 12 months after surgery
  Radiologic progression time following the RANO 2.0 criteria

SECONDARY OUTCOMES:
overall survival | 18 months after surgery
  patient survival time

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hwan Kim, MD, PhD, Principal Investigator — Department of Neurosurgery, Chungnam National University Hospital; Kijoon Yoon, PhD, Principal Investigator — Korea Advanced Institute of Science and Technology
Locations (1):
- Chungnam National University Hospital, Daejeon, Chungcheongnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No